CLINICAL TRIAL: NCT05003635
Title: External Vacuum Expansion: Evaluation in Breast Reconstructive Surgery
Brief Title: External Vacuum Expansion: Evaluation in Breast Reconstructive Surgery Evaluation in Breast Reconstructive Surgery
Acronym: EVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METC20-099
Record Dates: First submitted 2021-07-22; First posted 2021-08-12 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer Female
Keywords: fat grafting; lipoaspirate; fat injection; fat transfer; lipofilling; liposculpturing; lipoinjection; lipotransfer; breast reconstruction; external pre-expansion; BRAVA; EVE

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AFT+ EVEBRA device (intervention arm) (Active Comparator): Before and after the AFT surgery, patients are required to wear the EVEBRA expansion device for a total duration of 4 weeks. Thereafter patients will receive a PexyBra over the reconstructed breast.
  Pre-operatively patients are required to wear the device for a total of 200 hours.
  Interventions: Device: EVEBRA device
- AFT without EVEBRA device (control arm) (No Intervention): Patients will receive the AFT treatment for total reconstruction without the requirement of wearing the EVEBRA device.

INTERVENTIONS:
Device: EVEBRA device — Wear 2 weeks pre-operatively for a total duration of 200 hours. Wear 2 weeks post-operatively for 10 hours a day.
  Arms: AFT+ EVEBRA device (intervention arm)

SUMMARY:
This multicentre randomized controlled trial aims to evaluate a new breast reconstruction technique- autologous fat transfer (AFT). Female patients with breast cancer schedule to receive a mastectomy (or having undergone mastectomy in the past) will be randomized to undergo breast reconstruction with either AFT with the EVEBRA device(intervention group) or AFT without the EVEBRA device (control group). AFT will be evaluated in terms of volume, quality of life, aesthetic result, complications and oncological safety.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 23-69
* BMI 18-35 - stable weight, no fluctuations
* Have undergone a total mastectomy at least 3 months prior the study, whether therapeutic or prophylactic, whether unilateral or bilateral, with no resection of the pectoralis muscle
* Agrees to have reconstruction at the time of study involving only autologous fat grafting (AFT)
* Assessed by surgeon to have enough donor fat
* Passes a 20-minutes tolerance test with EVEBRA Device. (Patient will be fitted, instructed on the use, and given the EVEBRA Device to try in the office for 20 minutes. She passes if she tolerates its use, feels comfortable wearing it, and is able to comply with the required wear of the device.)

Exclusion Criteria:

* untreated breast cancer
* history of radiation therapy on the involved breast, even if it was part of a previous breast conservation procedure
* completed chemotherapy course less than 2 months prior (acceptable to still be on aromatase inhibitors)
* except for the biopsy leading to the diagnosis of cancer, had surgery to breast prior to the mastectomy (e.g., multiple biopsies, implant augmentation, mastopexy, fat grating)
* had mastectomy wound healing complications, e.g., seroma, wound breakdown, infection
* mastectomy defect/scar has significant skin excess and deep folds adherent to the chest wall
* has a pacemaker or aneurysm clips
* pregnancy or breastfeeding
* had a cardiac stent placed within the last 2 months
* claustrophobic, as reported by patient
* known current substance abuse, as reported by patient
* history of silicone allergy, as reported by patient
* history of Gadolinium allergy, as reported by patient
* history of lidocaine allergy, as reported by patient
* bleeding diathesis, whether primary or iatrogenic, as reported by patient cigarette smoker and/or Smokeless cigarette smokers, as reported by patient
* medical conditions that preclude breast reconstruction including uncontrolled hypertension or diabetes, renal failure, steroid dependent asthma, and on immuno- suppressant medications, as reported by patient

Ages: 23 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness measured in volume (MRI) | 1 year
  All women will have an MRI for Baseline Breast Volume measurement at the time of enrollment. Final breast volume will be also determined by MRI 6 months after the first grafting procedure (AFT#1).
  The primary effectiveness endpoint is the Percentage Augmentation of the mastectomy defect at 12 months after AFT#1.

SECONDARY OUTCOMES:
The quality of the reconstructed breast tissue as determined by MRI. | 12 months
  Presence + description of necrotic cysts (Scale: amount of cyst and size in centimeters)
The patient reported satisfaction at baseline and post-AFT using the Breast-Q Questionnaire | 12 months
  Qscore will be used to assess final scores. As described in the BREAST-Q Module, summed scores will be converted into a score from 0 (worst) to 100 (best) per domain. Higher scores reflect a better outcome.
Return of sensation to the breast as determined by Semmes-Weinstein monofilaments (map of the reconstructed breast mound with record of sensory levels) | 12 months
Visual/standard photographic appearance of the reconstructed breast will be determined using a Likert scale 1-5. | 12 months
  The aesthetic improvement will be rated using pre-operative and one year post-operative 2D images by a group of experts, breast cancer patients and age-matched male and female laymen. All parties rate the pre-/post- 3D images on a Likert scale (5 points) with one indicating no improvement and 5 indicating perfect improvement.
Difference in chest circumference between the peak of the reconstructed breast mound and the circumference just below the inframammary line | 12 months
  Difference noted in centimeters (cm)
Difference in bra cup size | 12 months
  Cup size before and after reconstruction will be noted .
Difference in Breast Volume from the randomization baseline after the three sessions of fat grafting (Final Reconstructed Breast Volumes) as measured by the validated Vectra 3D imaging system and the MRI. | 12 months
  Volume change will be noted in cubic centimetre(cc)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Piatkowski de Gryzmala, MD, MsC, Principal Investigator — Maastricht University Medical Center
Locations (3):
- Netherlands (3):
  - Maastricht University Medical Center+, Maastricht, Limburg
  - Amsterdam University Medical Center (VUMC), Amsterdam
  - Ziekenhuis groep Twente (ZGT), Hengelo